CLINICAL TRIAL: NCT04036851
Title: Peer Support to Mitigate the Impact of Stigma in Young HIV+ Pregnant & Postpartum Women: A Pilot Study
Brief Title: Peer Support to Mitigate the Impact of Stigma in Young HIV+ Pregnant & Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Professor Landon Myer, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 267/2019
Record Dates: First submitted 2019-07-16; First posted 2019-07-30 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local standard of care (No Intervention): Women receive integrated antenatal and HIV services during pregnancy and are referred to general adult HIV services after delivery; no standardized peer support groups exist for this patient population.
- Peer support intervention (Experimental): Women will be invited to attend monthly peer support groups during pregnancy and postpartum, separate from any routine health services.
  Interventions: Behavioral: Peer support intervention

INTERVENTIONS:
Behavioral: Peer support intervention — Peer support groups will meet monthly for the duration of follow-up, with separate groups for pregnant and postpartum women. Groups will be facilitated by women who are living with HIV and have experience of PMTCT services in this setting. Group sessions will include brief information and a structured discussion about a relevant topic, followed by opportunities for unstructured discussion.
  Arms: Peer support intervention

SUMMARY:
Young pregnant and postpartum women living with HIV are at the greatest risk of disengagement from HIV services and suboptimal adherence to antiretroviral therapy (ART). Among young women, stigma is a major barrier to retention in services and adherence to ART, and interventions are needed to combat stigma and improve ART outcomes. The investigators are conducting a pilot study of a peer support intervention to mitigate the negative effects of stigma in this population.

DETAILED DESCRIPTION:
Despite major reductions in mother-to-child HIV transmission (MTCT), young pregnant and postpartum women living with HIV remain a vulnerable group and experience the greatest risk of disengagement from services and suboptimal adherence to antiretroviral therapy (ART). HIV-related and intersectional stigmas are major barriers to uptake and retention in prevention of mother-to-child transmission (PMTCT) services and drive suboptimal adherence, and young women experience unique stigmas. Despite this, there are no evidence-based interventions to combat stigma and improve ART outcomes in this group. Peer support group interventions have shown promise in other populations, but have not been examined in young pregnant and postpartum women living with HIV. The investigators are conducting a pilot study of a peer support intervention to mitigate the negative effects of stigma in young pregnant and postpartum women living with HIV in South Africa. Participants will be allocated to the standard of care, in which no standardized peer support groups exist for this patient population, or to a peer support intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16-24 years
* Documented HIV infection
* Confirmed pregnant or recently postpartum
* Accessing antenatal or immediate postpartum PMTCT services at the study site
* Planning on remaining a resident of Cape Town for at least 6 months after enrolment
* Able to provide informed consent for research

Exclusion Criteria:

* Significant pre-existing psychiatric comorbidity that may impact ability to consent
* Stated intention to move outside of Cape Town during the 6 months after enrolment

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Retention and viral suppression | After 6 months of follow-up
  Combined endpoint of (i) retention in HIV services and (ii) HIV viral suppression. Women will be considered to have achieved the primary outcome if they are both retained in care and virally suppressed.

SECONDARY OUTCOMES:
Psychosocial outcomes | 6 months
  Psychosocial outcomes, including perceived social support and adherence self-efficacy, assessed using self-report questionnaires
Implementation of the intervention | 6 months
  Implementation of the peer support intervention including standardization, assessed using logs and process notes completed by counsellors who will deliver the intervention
Acceptability of the intervention | 6 months
  Acceptability of the peer support intervention, assessed as utilization and during in-depth interviews in a subset of participants
Health status | 6 months
  Maternal and infant health status, assessed using self-report and routine medical records
Health service use | 6 months
  Maternal and infant routine medical service use, assessed using self-report and routine medical records

CONTACTS AND LOCATIONS:
Overall Officials: Landon Myer, MBChB, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Gugulethu Community Health Centre, Cape Town, Western Cape, South Africa

REFERENCES:
- [Derived] Brittain K, Gomba Y, Noholoza S, Pellowski J, Mellins CA, Bekker LG, Kagee A, Remien RH, Abrams EJ, Myer L. HIV-related stigma, disclosure and social support: experiences among young pregnant and postpartum women living with HIV in South Africa. AIDS Care. 2023 Mar;35(3):399-405. doi: 10.1080/09540121.2022.2121957. Epub 2022 Sep 14. PMID 36102063